CLINICAL TRIAL: NCT03137836
Title: Effects of Sit-to-stand Desks on Behavior and Cognitive Function in Children
Brief Title: Classroom Standing Desks for Reducing Sitting Time in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Luís Bettencourt Sardinha, Full Professor, University of Lisbon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSardinha
Record Dates: First submitted 2016-09-13; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Sedentary Lifestyle; Cognitive Ability, General
MeSH Terms: conditions — Sedentary Behavior | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Sit-to-stand desks (Ergotron LearnFit®) will replace standard desks. In addition, meeting with parents and teacher's training will be conducted in order to support behavior change.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Control classroom will maintain their routine in sitting desks.

INTERVENTIONS:
Behavioral: Intervention — Multi-level intervention focused on school environment (furniture) will be conducted.
  Device: Sit-to-stand desks (Ergotron LearnFit®); Device: (Actigraph, Pensacola, FL, USA); Device: ActivPALTM .
  Arms: Intervention

SUMMARY:
In this trial the investigators aim to verify the potential impacts of a multi-level intervention with standing desks on behavior and cognitive function in children

DETAILED DESCRIPTION:
This is a cluster controlled trial conducted in a school setting. Two classes (intervention and control) of sixth grade will be selected from a large, centrally located school in Lisbon. The intervention will take place over a period of 16 weeks and will be composed of physical environmental (standing desks), social environment, and education/behavior components. Objective measurements of physical activity and sedentary behavior (ActiGraph GT3X+ accelerometer and activPAL inclinometer), school performance (students grades), attention (D2 test), memory (Rey complex figure), fluid intelligence (Raven's Progressive Matrices), visuo-spatial short term working memory (Corsi block-tapping test), processing speed and inhibitory function (Stoop test) will be assessed. Finally, anthropometry and stakeholders' perceptions will also be obtained at baseline and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 11 and 13 years-old
* Be able to postural changes

Exclusion Criteria:

* Do not return the written informed consent properly signed by parents/guardians

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-06-09 (Actual); Study Completion 2016-06-17 (Actual)

PRIMARY OUTCOMES:
Sedentary behavior | 16 weeks
  Sedentary behavior will be assessed trough the sitting time (min/day) given by ActivPALTM micro device (PAL Technologies Limited, Glasgow, UK). The device will be attached on anterior mid-line of the participants right thigh though 3MTM TegadermTM Transparent Film Roll (4 in x 11yd). Participants will wear the inclinometer continuously for seven days, including shower and sleep time, except in swimming activities. The ActivPAL3TM software v.7.2.32 will be used to data reduction. In addition to the baseline and follow-up measurements, the inclinometer will be used during the intervention just in school time to better clarify the sit-to-stand desks use.

SECONDARY OUTCOMES:
Physical activity | 16 weeks
  Physical activity will be measured though Actigraph GT3X+ accelerometers (Actigraph, Pensacola, FL, USA). Participants will be instructed to wear the device on the right rip (near the iliac crest) during waking hours for seven days. The device will be attached via an elastic belt and must will removed only in water-based activities. Will be considered a valid evaluations which had four or more days (including one of weekend) of a minimum of 600 minutes of wear. The Choi et al. [16] criteria of wear time and Evenson et al. [17] cuttoffs to PA intensities will be applicable with 15s epochs (collected at 30Hz) by Actilife v.6.10.4. The participants shall register in daily record the time which the device is removed and the reason.
Academic achievement | 16 weeks
  Participants grades will be obtained in both assessments points. Individual and sum of disciplines grades changes will be considered to comparisons purposes.
Participants self-reported measurements | 16 weeks
  Information about self-perception of physical and mental health, academic performance, behaviors (exercise and sleep habits) and social relationship will be assessed by a specific questionnaire for the participants. In addition, the intervention group ones will report their expectations (before) and perceptions (after) of the standing desks use.
Stakeholders perceptions | 16 weeks
  Parents/guardians (individual level) and teachers perceptions (cluster level) about discipline, social interaction, academic performance and health behaviors of the children will be collected by a questionnaire filled before and after the intervention.
Cost-effectiveness | 16 weeks
  Considering the costs of classroom environmental adaptations and their effects on primary and secondary outcomes, the incremental cost-effectiveness ratio will be calculated comparing with costs of a traditional classroom.
Cognitive function - Coop Corsi block-tapping test | 16 weeks
  Visual-spatial working memory capacity will be assessed through Coop Corsi block-tapping test. A 3 × 3 grid of 9 blocks indicates a spatial sequence by changing the colour of one block at a time, and participants were then asked to repeat that sequence by clicking on the blocks in the same order. During the 12 trials, sequence length increased by 1 block location each time the participant correctly repeated the sequence. Any error in repeating a sequence led to the next sequence being shortened by one location. The variable of interest was mean memory span, calculated as the average length of the three longest correctly repeated sequences.
Cognitive function - Stroop color test | 16 weeks
  Sensitivity to interference and the ability to suppress an automated response will be assessed using the Stroop color test. The Stroop test consists in two levels. Both levels involve the test word being placed in the center of the screen, with the target and distractor presented randomly on the right or left of the test word. The target position was counterbalanced for the left and right side within each test level. The participant is asked to respond as quickly as possible, using the left and right arrow keys, to identify the position of the target word. The variable of interest is the proportion of correct responses made.
Cognitive function - d2 test | 16 weeks
  Sustained attention and visual scanning ability will be assessed using the d2 test. This paper-and-pencil task requires participants to detect "d" symbols with two dashes (that may be located either both above, both below, or one above and one below the "d") among distractors ("d's" with one, three, or four marks or "p's" with one or two marks).
  The concentration performance score was determined on the number of correct responses minus errors. Higher scores indicate a better and more stable performance.
Neuropsychological assessment - Raven's matrices test | 16 weeks
  Neuropsychological assessment will be assessed using the Raven's Progressive Matrices. The test provides a simplified 36-item paper format. Each item contains a pattern problem with one part removed and six pictured inserts of which one contains the correct pattern. Participants point to the pattern piece they select or to its number. The total score is the total number of matrices completed correctly, and the test is thus scored out of 36.
Neuropsychological assessment - Rey-Osterrieth complex figure test | 16 weeks
  Neuropsychological assessment will be assessed using the Rey-Osterrieth complex figure test. The Rey-Osterrieth complex figure test (ROCF) is a neuropsychological assessment in which participants are asked to reproduce a complicated line drawing, first by copying it freehand (direct), and then drawing from memory (delayed copying). ROCF includes 18 units and the maximum score for each of the two tasks (direct and delayed copying) is 36. Two points are given when the element is correctly reproduced, 1 point when the reproduction is distorted, incomplete but placed properly, or complete but placed poorly; 0.5 point is credited when the element is distorted or incomplete and placed poorly. A zero score is given when the unit is absent or not recognizable.

CONTACTS AND LOCATIONS:
Overall Officials: Luís Sardinha, PhD, Study Chair — University of Lisbon
Locations (1):
- Danilo Rodrigues Pereira da Silva, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owen N. Sedentary behavior: understanding and influencing adults' prolonged sitting time. Prev Med. 2012 Dec;55(6):535-9. doi: 10.1016/j.ypmed.2012.08.024. Epub 2012 Sep 8. PMID 22968124
- [Background] Prince SA, Saunders TJ, Gresty K, Reid RD. A comparison of the effectiveness of physical activity and sedentary behaviour interventions in reducing sedentary time in adults: a systematic review and meta-analysis of controlled trials. Obes Rev. 2014 Nov;15(11):905-19. doi: 10.1111/obr.12215. Epub 2014 Aug 11. PMID 25112481
- [Background] Sedentary Behaviour Research Network. Letter to the editor: standardized use of the terms "sedentary" and "sedentary behaviours". Appl Physiol Nutr Metab. 2012 Jun;37(3):540-2. doi: 10.1139/h2012-024. Epub 2012 Apr 27. No abstract available. PMID 22540258
- [Background] Biswas A, Oh PI, Faulkner GE, Bajaj RR, Silver MA, Mitchell MS, Alter DA. Sedentary time and its association with risk for disease incidence, mortality, and hospitalization in adults: a systematic review and meta-analysis. Ann Intern Med. 2015 Jan 20;162(2):123-32. doi: 10.7326/M14-1651. PMID 25599350
- [Background] Owen N, Sugiyama T, Eakin EE, Gardiner PA, Tremblay MS, Sallis JF. Adults' sedentary behavior determinants and interventions. Am J Prev Med. 2011 Aug;41(2):189-96. doi: 10.1016/j.amepre.2011.05.013. PMID 21767727
- [Background] Tremblay MS, LeBlanc AG, Kho ME, Saunders TJ, Larouche R, Colley RC, Goldfield G, Connor Gorber S. Systematic review of sedentary behaviour and health indicators in school-aged children and youth. Int J Behav Nutr Phys Act. 2011 Sep 21;8:98. doi: 10.1186/1479-5868-8-98. PMID 21936895
- [Background] Ridgers ND, Salmon J, Ridley K, O'Connell E, Arundell L, Timperio A. Agreement between activPAL and ActiGraph for assessing children's sedentary time. Int J Behav Nutr Phys Act. 2012 Feb 19;9:15. doi: 10.1186/1479-5868-9-15. PMID 22340137
- [Background] Clemes SA, Barber SE, Bingham DD, Ridgers ND, Fletcher E, Pearson N, Salmon J, Dunstan DW. Reducing children's classroom sitting time using sit-to-stand desks: findings from pilot studies in UK and Australian primary schools. J Public Health (Oxf). 2016 Sep;38(3):526-533. doi: 10.1093/pubmed/fdv084. Epub 2015 Jun 14. PMID 26076699
- [Background] Gardner B, Smith L, Lorencatto F, Hamer M, Biddle SJ. How to reduce sitting time? A review of behaviour change strategies used in sedentary behaviour reduction interventions among adults. Health Psychol Rev. 2016;10(1):89-112. doi: 10.1080/17437199.2015.1082146. Epub 2015 Sep 16. PMID 26315814
- [Background] Benden ME, Blake JJ, Wendel ML, Huber JC Jr. The impact of stand-biased desks in classrooms on calorie expenditure in children. Am J Public Health. 2011 Aug;101(8):1433-6. doi: 10.2105/AJPH.2010.300072. Epub 2011 Mar 18. PMID 21421945
- [Background] Hinckson E, Salmon J, Benden M, Clemes SA, Sudholz B, Barber SE, Aminian S, Ridgers ND. Standing Classrooms: Research and Lessons Learned from Around the World. Sports Med. 2016 Jul;46(7):977-87. doi: 10.1007/s40279-015-0436-2. PMID 26626071
- [Background] Minges KE, Chao AM, Irwin ML, Owen N, Park C, Whittemore R, Salmon J. Classroom Standing Desks and Sedentary Behavior: A Systematic Review. Pediatrics. 2016 Feb;137(2):e20153087. doi: 10.1542/peds.2015-3087. Epub 2016 Jan 22. PMID 26801914
- [Background] Mirwald RL, Baxter-Jones AD, Bailey DA, Beunen GP. An assessment of maturity from anthropometric measurements. Med Sci Sports Exerc. 2002 Apr;34(4):689-94. doi: 10.1097/00005768-200204000-00020. PMID 11932580
- [Background] Choi L, Liu Z, Matthews CE, Buchowski MS. Validation of accelerometer wear and nonwear time classification algorithm. Med Sci Sports Exerc. 2011 Feb;43(2):357-64. doi: 10.1249/MSS.0b013e3181ed61a3. PMID 20581716
- [Background] Evenson KR, Catellier DJ, Gill K, Ondrak KS, McMurray RG. Calibration of two objective measures of physical activity for children. J Sports Sci. 2008 Dec;26(14):1557-65. doi: 10.1080/02640410802334196. PMID 18949660
- [Derived] Silva DR, Machado DGS, Pinto F, Judice PB, Minderico CS, Collings PJ, Cyrino ES, Sardinha LB. Effect of a 16-week multi-level classroom standing desk intervention on cognitive performance and academic achievement in adolescents. Sci Rep. 2022 Sep 1;12(1):14504. doi: 10.1038/s41598-022-18248-y. PMID 36050353